CLINICAL TRIAL: NCT04199650
Title: Definition of Acute Respiratory Distress Syndrome in Plateau of Qinghai in China: Verification of Berlin Definition Plateau Criteria
Brief Title: Definition of ARDS in Qinghai Province: Verification of Berlin Definition Plateau Criteria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Collaborators: Affiliated Hospital of Qinghai University (Other)
Responsible Party: Principal Investigator, Chun Pan, Deputy chief physician, Southeast University, China
Other Study IDs: ARDS Plateau Criteria
Record Dates: First submitted 2019-12-05; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: ARDS; High Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild ARDS: 153mmHg<PaO2/FiO2≤230mmHg
- Moderate ARDS: 76mmHg<PaO2/FiO2≤153mmHg
- Severe ARDS: PaO2/FiO2≤76mmHg

SUMMARY:
The severity stratification criteria for acute respiratory distress syndrome (ARDS) in Xi'ning Qinghai province (mean altitude: 2200m) were clarified according to the oxygenation index (PaO2/FiO2).

DETAILED DESCRIPTION:
This study is a single-center retrospective study. According to the Berlin diagnostic standard, ARDS patients admitted to the Department of severe Medicine, affiliated Hospital of Qinghai University from January 2018 to December 2018 were divided into three groups: mild (153mmHg < PaO2/ FiO2 ≥ 230 mmHg), moderate (76mmHg < PaO2/ FiO2 ≥ 153 mmHg) and severe (PaO2/ FiO2 ≥ 76 mmHg). The ICU mortality, 28-day mortality, non-ventilator time in ICU, ICU hospitalization time and non-I hospitalization were observed respectively. The difference of CU time and total hospitalization days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Meet the diagnostic criteria of ARDS
* Receive invasive mechanical ventilation

Exclusion Criteria:

* Receive a large number of hormone shock therapy in a short period of time
* Death within a short period of time (< 24 h) after mechanical ventilation
* No chest imaging data
* Data missing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2018 to December 2018, patients admitted to the department of critical care, affiliated hospital of qinghai university were diagnosed with acute respiratory distress syndrome according to Berlin Definition.
Sampling Method: Non-Probability Sample
Enrollment: 253 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-01-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | up to 24 weeks
  Mortality during treatment in ICU
28-days mortality rate | 28 days after discharge
  Mortality at 28 days of hospitalization

SECONDARY OUTCOMES:
Ventilator Free time | up to 24 weeks
  Ventilator time not used in ICU
Ventilator time | up to 24 weeks
  Ventilator time in ICU
Hospital length of stay | up to 24 weeks
  Total length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Liu Xiaoqin, Bachelor, Principal Investigator — Affiliated Hospital of Qinghai University
Locations (1):
- ChunPan, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Liu X, Pan C, Si L, Tong S, Niu Y, Qiu H, Gan G. Definition of Acute Respiratory Distress Syndrome on the Plateau of Xining, Qinghai: A Verification of the Berlin Definition Altitude-PaO2/FiO2-Corrected Criteria. Front Med (Lausanne). 2022 Feb 23;9:648835. doi: 10.3389/fmed.2022.648835. eCollection 2022. PMID 35280910